CLINICAL TRIAL: NCT06159127
Title: Self-Management Assistance for Recommended Treatment (SMART)@Home Care
Brief Title: SMART@Home Feasibility Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMART@Home
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Asthma; Asthma in Children
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART@Home (Experimental): Use of the SMART@Home app for medication and symptom tracking, spirometry feedback
  Interventions: Behavioral: SMART@Home
- Control (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: SMART@Home — Daily medication and diary completion reminders are provided to participants. Additional educational content regarding self-management skills will be provided.
  Arms: SMART@Home

SUMMARY:
The proposed research addresses the limitations or lack of a digital platform to provide remote care of medically complex patients. Previous attempts have had poor clinical validity and suffered lack of patient engagement. The study team will deconstruct the previously implemented SMART platforms to create a roadmap, platform, and template to guide clinicians to create new tools.

Results from Phase 1 of this project highlighted the need for connectivity between the SMART@Home app and Bluetooth-enable devices to provide objective disease activity data as well as integration with Epic electronic health record so that providers can use the data to inform treatment planning and decision making. A subsequent pilot user validation trial is also needed to confirm development goals were met. Conducting a pilot user validation trial of the SMART@Home asthma tracker, spirometer, and action plan is the purpose of the next phases of this study.

A beta test the SMART@Home Asthma Tracker and asthma action plan algorithm will take place with approximately 8 participants. Beta testing will have participants record simulated increases in symptoms to ensure appropriate levels of care is communicated via the app. Then, a group of 40 adolescent (ages 12-17) patients with asthma for a 6-month pilot Randomized Control Trial (RCT). Participants will be randomized into either the IMAAP SMART@Home (n=20) or control (n=20) groups following the completion of baseline measures to test the interactive asthma action plan functionality and impact.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a chronic medical condition requiring regular treatment, i.e., asthma
* Ages 12-18
* English fluency for patient and caregiver

Exclusion Criteria:

* Diagnosis of pervasive developmental disorder in patient or caregiver as determined by medical chart review
* Diagnosis of serious mental illness (e.g., schizophrenia) in patient or caregiver as determined by medical chart review

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | 6 months
  Monthly adherence will be calculated by comparing doses taken to doses recommended by IMAAP. Participants will also report rescue medication use each month when completing the ACT.
Number of days app used | 6 months
  Number of diaries completed by participant

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hommel, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Rachelle Ramsey, PhD, Study Chair — Children's Hospital Medical Center, Cincinnati; Matt Wortman, PhD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States